CLINICAL TRIAL: NCT05557838
Title: An Open-label, Multi-center Phase IIIb Study of Durvalumab and Tremelimumab as First-Line Treatment in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Study of Durvalumab Plus Tremelimumab as First-line Treatment in Chinese Patients With Unresectable Hepatocellular Carinoma
Acronym: TREMENDOUS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D419CR00026
Record Dates: First submitted 2022-09-14; First posted 2022-09-28 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cohort 1 (Experimental): durvalumab in combination with tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- cohort 2 (Experimental): durvalumab in combination with tremelimumab
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous infusion)
  Other Names: MEDI4736
Drug: Tremelimumab — Tremelimumab IV (intravenous infusion)

SUMMARY:
This is a prospective, open label, multi-center, interventional study to assess the safety and efficacy of Druvalumab plus Tremelimumab as first-line treatment in Chinese patients with unresectable hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HCC based on histopathological findings from tumor tissue or radiologically findings
* No prior systemic therapy for HCC
* Barcelona Clinic Liver Cancer (BCLC) stage B (not eligible for locoregional therapy) or stage C
* Child-Pugh Score class A or B
* ECOG performance status (PS) of 0-2 at enrollment (Child-Pugh Score class A and ECOG PS of 0-1 will be enrolled in cohort 1 and Child-Pugh Score class B or ECOG PS of 2 will be enrolled in cohort 2)
* At least 1 measurable lesion per RECSIT 1.1 guidelines

Exclusion Criteria:

* Hepatic encephalopathy within past 12 months or requirement for medication to prevent or control encephalopathy
* Clinically meaningful ascites
* Main portal vein tumor thrombosis
* Active or prior documented GI bleeding (eg, esophageal varices or ulcer bleeding) within 6 months
* HBV and HVC co-infection, or HBV and Hep D co-infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
≥Grade 3 Adverse Events and Adverse Events of Special Interest of Cohort 1 | From the time of signature of informed consent, throughout the treatment period, and up to the follow-up period, assessed up to 29 months

SECONDARY OUTCOMES:
≥Grade 3 Adverse Events and Adverse Events of Special Interest of Cohort 2 | From the time of signature of informed consent, throughout the treatment period, and up to the follow-up period, assessed up to 29 months
Overall Survival (OS) | From the first dose of treatment to the date of death, regardless of the actual cause of the subject's death, assessed up to 29 months
Progression Free Survival (PFS) per RECIST v1.1/mRECIST | From first dose of treatment until progression per RECIST 1.1/ mRECIST as assessed by the Investigator or death due to any cause prior to progression, assessed up to 15 months
Objective Response Rate (ORR) per RECIST 1.1/ mRECIST | Until progression, assessed up to 15 months
Disease Control Rate (DCR) per RECIST 1.1/ mRECIST | Until progression, assessed up to 15 months
Rate of Adverse Events | From the time of signature of informed consent, throughout the treatment period, and up to the follow-up period, assessed up to 29 months
Duration of response (DoR) per RECIST 1.1/mRECIST | From the first dose, until progression, assessed up to 15 months

CONTACTS AND LOCATIONS:
Locations (18):
- China (18):
  - Research Site, Beijing
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhangjiagang
  - Research Site, Zhengzhou

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient- level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  Plan Description: All request will be evaluated as per the Az disclosure commitment:
  https://astrazenecaarouptrials.pharmacm.com/ST/Submission/Disclosure Yes. indicates that Az are accepting requests for IPD ,but this does not mean are quests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitment at made to the EFPIA Pharma Data Sharing Principles .For details of our timeline please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool.
  Signed Data Sharing Agreement(non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to a air access. For additional details. please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home